CLINICAL TRIAL: NCT06835777
Title: Neurophysiological Mechanisms of Placebo and Nocebo Effects in Sports - Protocol Paper of a Randomised Controlled Study
Brief Title: Neurophysiological Mechanisms of Placebo and Nocebo Effects in Sports - a Protocol Paper
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Principal Investigator, Janina Hanssen, PhD Candidate, Canterbury Christ Church University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ETH2324-0198
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Placebo Effect; Nocebo Effect
Keywords: EEG; Placebo; Nocebo; Sports Performance

STUDY DESIGN:
Intervention Model Description: randomised controlled trail, four parallel arms (positive-expectations, negative-expectations, control , natural history)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- positive-expectations (Experimental): The positive-expectations intervention will consist of two inert pills filled with cornstarch and a manipulation of beliefs regarding the given substance and it's effects. Participants will be informed that the inert pills are neurostimulants, usually used in the context of depression and other mental health issues and that they can positively affect sports performance. Participants will be reinforced about these effects throughout testing via implicit adjectives regarding potential sensations they might experience after pill intake. Reinforcement of beliefs and subsequent strength testing will be EEG controlled.
  Interventions: Combination Product: Positive Expectation
- negative-expectations (Experimental): The negative-expectations intervention will consist of two inert pills filled with cornstarch and a manipulation of beliefs regarding the given substance and it's effects. Participants will be informed that the inert pills are neuro-depressants, which relieve anxiety and can negatively affect sports performance. Participants will be reinforced about these effects throughout testing via implicit adjectives regarding potential sensations they might experience after pill intake. Reinforcement of beliefs and subsequent strength testing on day two will be EEG controlled.
  Interventions: Combination Product: Negative Expectation
- control (Active Comparator): The control intervention consists of the same testing procedure as the other intervention groups, but no pills or manipulation of beliefs will be administered. Participants will be given a neutral presentation on the testing procedure of the isometric strength testing. Neutral adjectives will be presented instead of a reinforcement of beliefs. Presentation of adjectives and subsequent strength testing will be EEG controlled.
  Interventions: Other: Control
- natural history (No Intervention): Participants will neither receive an EEG nor any sort of intervention. They will do the isometric strength testing on two different occasions like the other groups and will not receive any sort of manipulation of beliefs.

INTERVENTIONS:
Combination Product: Positive Expectation — The lead researcher will deliver a short presentation (8 minutes) to participants informing them about the deceptive substance, presenting it as a performance enhancing neurostimulant,. Participants will be given the opportunity to ask questions and will receive a handout of the key points of the presentation. After the presentation, participants will be set up with a high-density EEG and given two inert pills filled with cornstarch. Participants will be reminded of the performance enhancing qualities of the deceptive substance by implicit adjectives on a screen. Afterwards, experimental performance outcomes will be collected using a dynamometer.
  Arms: positive-expectations
Combination Product: Negative Expectation — The lead researcher will deliver a short presentation (8 minutes) to participants informing them about the deceptive substance, presenting it as a performance inhibiting neuro-depressant. Participants will be given the opportunity to ask questions and will receive a handout of the key points of the presentation. After the presentation, participants will be set up with a high-density EEG and given two inert pills filled with cornstarch. Participants will be reminded of the performance inhibiting qualities of the deceptive substance by implicit adjectives on a screen. Afterwards, experimental performance outcomes will be collected using a dynamometer.
  Arms: negative-expectations
Other: Control — The lead researcher will deliver a short presentation (8 minutes) to participants informing them about EEG research and set ups and give general information about isometric strength testing. They will be shown neutral adjectives unrelated to performance instead of implicit adjectives related to performance (experimental groups). EEG set up and strength testing remains the same as the experimental groups.
  Arms: control

SUMMARY:
This clinical trial aims to investigate the neurophysiological mechanisms of placebo and nocebo effects on sports performance, using Electroencephalography (EEG) and isometric strength testing of the lower extremities.

The primary objective of this trial is to identify temporal mechanisms and cortical regions and networks involved in generating placebo and nocebo effects before (expectation) and at onset of athletic performance (perception).

The trial will include four groups, two of them experimental, one an active control and one natural history, meaning participants in this group will receive no intervention and won't be EEG controlled. Data will be collected on two occasions with baseline data for EEG, expectations and performance as well as key participant characteristics being collected on day one. On day two, in a deceptive process, participants in the two experimental groups will take an inert substance presented as either performance enhancing or inhibiting and subsequently experience a reinforcement of beliefs via exposure to explicit adjectives. EEG data will be collected during reinforcement of beliefs. In the active control group, participants will receive no substance, but this group will follow the same procedure as the experimental groups with neutral adjectives. Participants will then perform isometric strength and fatigue resistance tests on an isometric dynamometer. EEG data as well as subjective data on expectations and rating of perceived exhaustion will be collected.

DETAILED DESCRIPTION:
This trial will examine temporal and spatial aspects of neurophysiological mechanisms behind nocebo and placebo effects before (expectation) and at exercise onset (perception) using high-density EEG. It will further investigate possible predictors of responsiveness and non-responsiveness to acute placebo and nocebo stimuli in the context of sports, notably interpretating psychological mechanisms (e.g. personality, beliefs, expectations) as well as temporal neurophysiological measures.

This study is designed as a randomized, controlled clinical trial (RCT) with data collection on two different occasions and four parallel groups: 1) positive-expectations, 2) negative-expectations, 3) control, and 4) natural history.

The first three groups will be addressed as intervention groups. On the first visit, participants' baseline data, specifically performance measures (all groups) and EEG data (all but natural history), as well as key characteristics will be collected. On the second visit, in the belief groups, participants will receive an in-person manipulation of beliefs and two placebo pills and will be informed that they are expected to positively (positive-expectations) or negatively (negative-expectations) affect their isometric strength and fatigue resistance measured using a Biodex System 4 Isokinetic Dynamometer in a 5x5sec test protocol with a minimum of 1 minute rest in between sets. In addition, after a resting period of three minutes, they will perform an isometric knee extension hold to failure at 60% MVC. The control group and the natural history group will receive no pills, with the control group receiving a neutral explanation of EEG data, its relevance and general information about isometric strength testing and the natural history group not receiving EEG at all, but serving as a control to the potential influence of experiencing an EEG set up on performance measures. The primary endpoints of this trial are placebo and nocebo induced changes in EEG signaling via Event Related Potentials (ERPs) during administration of reinforcements of beliefs through words as well as during expectancy and perception phases of physical performance.

The key question of this trial is whether participants exposed to placebo or nocebo stimuli will exhibit distinct neural activity pattern (temporal and spatial) in the context of sports performance. The second major question is, whether individual differences in character traits and states as well as motivation and beliefs can significantly predict the magnitude or likeliness of placebo and nocebo responses in participants' performance in an isometric strength and fatigue resistance task. In addition, EEG data to better understand the valence of and emotional response to words will be used to further investigate how semantics and our choice of words influence susceptibility to placebo and nocebo effects in other people. Several elements that were not adequately addressed in previous studies will be incorporated into this RCT:

(1) temporal and spatial aspects of neural correlates of placebo and nocebo effects in sports, (2) hard data (EEG) on how an individual reacts to semantic implications on performance and (3) correlation of subjective ratings of expectations of performance and data from neural processes associated with affective processing, emotional valence and motivation (LPP,LPC) and anticipation as well as motor preparation (CNV). To further understand the above point may result in a change on how athletes, coaches and therapists approach placebo and nocebo effects in the context of sports performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants (18+)
* physically active (WHO, 2020)
* no medical history pf psychological disorders/mental health issues
* no acute or regular medication intake
* no severe injury to the lower limb within the last 6 months
* proficient in english
* normal or corrected eyesight

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG data - performance | From collection of baseline data on day one to the end of day two of data collection.
  Temporal neurophysiological data measured by EEG. The Continuous Negative Variation (CNV), an Event Related Potential (ERP), will be used to differentiate positive and negative expectations as well as motor preparation before and at onset of isometric strength testing.
EEG data - reinforcement of beliefs | From collection of baseline data on day one to the end of day two of data collection.
  Event related potentials (ERP) will be investigated during the reinforcement of beliefs, specifically the late positive potential (LPP) and the late positive component (LPC).
EEG, exploratory source analysis | From collection of baseline data on day one to the end of day two of data collection
  In addition to ERP data, Low-Resolution Electromagnetic Tomography (LORETA) will be used in an exploratory approach to identify specific neural origins associated with placebo and nocebo responses.

SECONDARY OUTCOMES:
Performance Output, Isometric Forces | From collection of baseline data on day one to the end of day two of data collection.
  Peak Isometric Force: Measured in Newton-meters (Nm) as the maximum force output during a 5-second unilateral knee extension contraction.
  Average Isometric Force: Calculated as the mean force output in Nm maintained over a 5-second unilateral knee extension contraction.
  Isometric Force output data will be analysed in a within and between analysis, the latter being normalized to body mass (Nm/kg).
Performance Output, Force Consistency | From collection of baseline data on day one to the end of day two of data collection.
  Force Consistency:
  Assessed by comparing peak and average force outputs in Nm across five consecutive trials of 5-second contractions.
Performance Output, Endurance Hold and Fatigue Resistance | From collection of baseline data on day one to the end of day two of data collection.
  Fatigue Resistance and Endurance Hold:
  Evaluating the time to failure at the 60% maximally voluntary contraction (MVC) hold.
Performance Output, Recovery Capacity | From collection of baseline data on day one to the end of day two of data collection.
  Recovery Capacity:
  Determined by examining the ability to maintain force output in Nm across trials with 1-minute rest intervals between contractions.
Heartrate | From collection of baseline data on day one to the end of day two of data collection.
  Heartrate (bpm) will be collected during and before physical performance as well as during EEG data collection.
Rate of Perceived Exertion (RPE) | From collection of baseline data on day one to the end of day two of data collection.
  Rate of perceived exertion (RPE) will be used to assess subjective effort and closeness to failure after isometric strength testing
Electromyographic (EMG) Data | From collection of baseline data on day one to the end of day two of data collection.
  EMG data of the M. vastus lateralis of the dominant leg during isometric performance tests will be collected.

OTHER OUTCOMES:
Questionnaires - Anxiety | From collection of baseline data on day one to the end of day two of data collection.
  Further outcomes measures include questionnaires and inventories to assess key personality traits and states, motivation and beliefs.
  1. Cognitive and Somatic State Anxiety levels measured by the Competitive Sport Anxiety Inventory-2 (CSAI-2).
Questionnaires - Motivation and Perception of Ability | From collection of baseline data on day one to the end of day two of data collection.
  A 7-point Likert scale will be used to assess the participants' achievement motivation and their approach to performance.
Questionnaires - Optimism | From collection of baseline data on day one to the end of day two of data collection.
  We will use the Life Orientation Test-Revised (LOT-R) to test for the level of optimism versus pessimism.
Questionnaires - Sport supplement use and belief | From collection of baseline data on day one to the end of day two of data collection.
  We will collect data on participants' use of and beliefs on sport supplements.
Questionnaires - Resilience | From collection of baseline data on day one to the end of day two of data collection.
  Participants' beliefs about their own general resilience will be assessed using the Resilience Evaluation Scale (RES).
Questionnaires - Sensitivity | From collection of baseline data on day one to the end of day two of data collection.
  We will assess participants' sensitivity to internal bodily sensations using the Body Vigilance Scale (BVS).
Questionnaires - Emotions | From collection of baseline data on day one to the end of day two of data collection.
  Positive and negative affects will be measured before data collection and after pill administration using a modified version of the Positive and Negative Affect Schedule (PANAS) using the subscales investigating negative affect, positive affect, fear, self-assurance, attentiveness and fatigue.
Questionnaires - Expectations of performance | From collection of baseline data on day one to the end of day two of data collection.
  We will assess pre- and post-intervention expectancy/perception levels of performance as well as the participants' expectancies and perceptions of substance effect before and after data collection using a 10 point Visual Analogue Scale (VAS) and 7 point Likert scale respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Canterbury Christ Church University, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No